CLINICAL TRIAL: NCT06384469
Title: The Impact of Rhinoplasty Approach and Used Autologous Cartilage Grafts on the Nasal Skin-soft Tissue Envelope Metabolism
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital Sestre Milosrdnice (Other)
Responsible Party: Principal Investigator, Mateo Čukman, medical doctor, resident, University Hospital Sestre Milosrdnice
Other Study IDs: 98984697615
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Rhinoplasty; Nasal Skin-soft Tissue Envelope Metabolism; Lactic Acid; Autologous Cartilage Grafting
Keywords: Open rhinoplasty approach; Closed rhinoplasty approach; Lactic acid; Skin-soft tissue envelope; Metabolism; Autologous cartilage grafting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients undergoing open rhinoplasty approach: Patients undergoing open rhinoplasty approach, of which most of will be augmented by using autologous cartilage grafts.
- Patients undergoing closed approach rhinoplasty.: Patients undergoing closed approach rhinoplasty of which only few will be augmented by using autologous cartilage grafts.

SUMMARY:
This is a prospective observation cohort investigation. Patients, that is participants, undergoing primary functional rhinoplasty will be evaluated in terms of measuring capillary blood lactic acid concentration in the nasal skin-soft tissue envelope immediately after the procedure and 7 days after the procedure.

The aim of our study is to test whether or not different rhinoplasty approaches and volume of the used autologous cartilage grafts impact the nasal skin-soft tissue metabolism.

DETAILED DESCRIPTION:
This is a prospective observation cohort investigation.100 adult participants undergoing primary functional rhinoplasty between the January 2nd 2025 and January 2nd 2026 will be assessed in terms of measuring capillary blood lactic acid concentration in the nasal skin-soft tissue envelope immediately after the procedure and 7 days after the procedure. Prior to conducting the investigation, the participants will need to sign an informed consent for participating in the study, which would be previously approved by the ethics committee. For measuring capillary blood lactic acid concentration investigators are to use StatStrip® Lactate device and test strips. The volume of the used autologous cartilage autografts will be measured as well by using the water displacement method. Other used information regarding demographics and operation details will be drawn from the hospital's information systems, to which only medical personnel has an access. Using statistical analysis investigators are to perform the independent samples t-test, that is the Mann-Whitney U test, to analyze whether or not there is a difference in lactic acid concentration in participants undergoing open vs closed rhinoplasty approach. Furthermore by using Person's correlation coefficient method, the correlation between the used autologous cartilage grafts volume and lactate concentration will be assessed. The results of the lactic acid concentration will be interpreted with an assistance of the medical biochemistry and laboratory medicine specialist.

The aim of our study is to test whether or not different rhinoplasty approaches and volume of the used autologous cartilage grafts impact the nasal skin-soft tissue metabolism.

Since the investigation is to be performed during the regular working hours and since there is no intervention, no external funding will be necessary.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing primary functional rhinoplasty who comply with the study
* Adult patients undergoing primary functional rhinoplasty who have singed the informed consent, previously approved by the ethics commitee.

Exclusion Criteria: -

* patients with previous surgical procedures to the nose
* patients with greater previous injury or burns to the nasal skin
* patients with autoimmune skin conditions
* patients with significant cardiovascular diseases
* patients unwilling to comply with the study
* patients who do not want to sign the informed consent, previously approved by the ethics commitee.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients between 18 and 80 years of age, scheduled for primary functional rhinoplasty, who are willing to comply with the study and sign the informed consent, previously approved by the ethics commitee.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-02 (Estimated); Primary Completion 2026-01-02 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Difference of capillary blood lactic acid concentration in the nasal skin-soft tissue envelope depending on the rhinoplasty approach | immediately after the surgical procedure and 7 days after the procedure
  In participants undergoing primary functional rhinoplasty, the capillary blood lactic acid concentration from the skin-soft tissue envelope will be assessed by using Statstrip lactate measuring device and Statstrip test strips immediately after the procedure and 7 days after the procedure.
Correlation between the used autologous cartilage graft volume and lactic acid concentration in the nasal skin-soft tissue envelope | immediately after the surgical procedure and 7 days after the procedure
  In the same participants undergoing different rhinoplasty approach, the volume of the used autologous cartilage grafts will be measured by using water displacement method, and this result will be correlated with the capillary blood lactic acid concentration from the skin-soft tissue envelope.

CONTACTS AND LOCATIONS:
Overall Officials: Marko Velimir Grgić, MD, PhD, Study Chair — UHC Sestre milosrdnice

IPD SHARING:
Plan to Share IPD: No
Individual participant data are not to be shared with other researchers.